CLINICAL TRIAL: NCT06994949
Title: Assessing CSF Flow Dynamics in Pediatric Hemorrhagic Hydrocephalus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eva Sevick (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Eva Sevick, Professor, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-21-0809; R01NS126437 (NIH)
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Post-hemorrhagic Hydrocephalus (PHH)
Keywords: cerebrospinal fluid (CSF); premature infants; indocyanine green (ICG)
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- fCTOT and NIRF imaging with ICG (Experimental)
  Interventions: Device: fCTOT cap; Device: NIRF planar imaging; Drug: ICG

INTERVENTIONS:
Device: fCTOT cap — The fCTOT cap will be placed on the infant's head . After the MRI, fiber optics will be connected to the cap while donned on the infant and measurements will commence. After initial CSF diversion, a 0.5 cc volume of ICG solution will injected into the subcutaneous reservoir and measurements will be conducted using the fCTOT for 30 minutes. The fCTOT cap will be removed and NIRF planar imaging will be conducted to detect ICG in the subarachnoid space (SAS), draining cervical lymph nodes, along the spinal canal, and in the abdomen, where liver signals are expected. The infant will be transported back to the ICU where CSF diversion will continue and daily, 30 minutes NIRF imaging sessions may be conducted to detect ventricular flow into the SAS and liver clearance. Daily NIRF imaging will be performed in the neonatal intensive care unit (NICU) for as long as 7 days or until the ICG has cleared from the body from liver and/or CSF diversion.
Device: NIRF planar imaging — The fCTOT cap will be placed on the infant's head . After the MRI, fiber optics will be connected to the cap while donned on the infant and measurements will commence. After initial CSF diversion, a 0.5 cc volume of ICG solution will injected into the subcutaneous reservoir and measurements will be conducted using the fCTOT for 30 minutes. The fCTOT cap will be removed and NIRF planar imaging will be conducted to detect ICG in the SAS, draining cervical lymph nodes, along the spinal canal, and in the abdomen, where liver signals are expected. The infant will be transported back to the ICU where CSF diversion will continue and daily, 30 minutes NIRF imaging sessions may be conducted to detect ventricular flow into the SAS and liver clearance. Daily NIRF imaging will be performed in the NICU for as long as 7 days or until the ICG has cleared from the body from liver and/or CSF diversion.
Drug: ICG — The fCTOT cap will be placed on the infant's head . After the MRI, fiber optics will be connected to the cap while donned on the infant and measurements will commence. After initial CSF diversion, a 0.5 cc volume of ICG solution will injected into the subcutaneous reservoir and measurements will be conducted using the fCTOT for 30 minutes. The fCTOT cap will be removed and NIRF planar imaging will be conducted to detect ICG in the SAS, draining cervical lymph nodes, along the spinal canal, and in the abdomen, where liver signals are expected. The infant will be transported back to the ICU where CSF diversion will continue and daily, 30 minutes NIRF imaging sessions may be conducted to detect ventricular flow into the SAS and liver clearance. Daily NIRF imaging will be performed in the NICU for as long as 7 days or until the ICG has cleared from the body from liver and/or CSF diversion.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ventricular microdosing of indocyanine green (ICG) in order to assess cerebrospinal fluid (CSF) ventricular dynamics and extracranial CSF outflow using fluorescent Cap-based Transcranial Optical Tomography (fCTOT) and Near-InfraRed Fluorescent (NIRF) imaging and to evaluate inflammation markers of the CSF and to correlate with CSF ventricular dynamics, extracranial outflow into the lymphatics, ventriculomegaly, and patient's clinical outcome in order to understand how inflammation may impact that status of extracranial outflow.

ELIGIBILITY:
Inclusion Criteria:

* Children born premature currently in the NICU with a diagnosis of PHH who have undergone ventricular reservoir placement.
* For the first four study subjects, we will attempt for the child to undergo CT cisternography when clinically stable 3-4 weeks after reservoir placement.

Exclusion Criteria:

* Parents who do not consent for procedure on their child
* Children who are deemed clinically unstable or unsuitable for imaging by clinical staff as defined by the subject's level of intensive care (e.g. can the subject be repositioned without compromise to the level of care needed or condition)
* Children known or suspected to have allergy to iodine or ICG
* Children who do not have a subcutaneous reservoir for CSF diversion from the lateral ventricle

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2029-01-03 (Estimated); Study Completion 2029-01-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants 1-2 weeks of age who present with continuing ventriculomegaly after CSF diversion as assessed by the clinical MRI examination | end of study (about 10 days form baseline)
Number of participants 1-2 months of age who present with elevated ventriculomegaly after Endoscopic Third Ventriculostomy (ETV)/Choroid Plexus Cauterization (CPC) as assessed by the clinical MRI examination | end of study (about 10 days form baseline)
Number of participants 1-6 months of age who present with continuing ventriculomegaly after ETV/CPC as assessed by the clinical MRI examination | end of study (about 10 days form baseline)

SECONDARY OUTCOMES:
Amount of pro-inflammatory cytokines measured in pg/ml | end of study (about 10 days form baseline)
  Cytokines include Interleukin (IL)-1beta IL-4 IL-6 IL-10 IFNgamma TNFalpha Neural Cell Adhesion Molecule 1 (NCAM-1) Monocyte chemoattractant protein-1(MCP-1) IL-18

CONTACTS AND LOCATIONS:
Overall Officials: Manish Shah, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No